CLINICAL TRIAL: NCT02880995
Title: Positron Emission Tomography(PET) With 3,4-dihydroxy-6-18-fluoro-l-phenylalanine ([18 Fluorine(F)]DOPA) Determinants and Predictors of Treatment Response in Psychosis
Brief Title: [18 Fluorine(F)]DOPA Determinants and Predictors of Treatment Response in Psychosis
Acronym: DPTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Euitae Kim, professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOPAPET_predictor-1000
Record Dates: First submitted 2016-08-04; First posted 2016-08-26 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
Keywords: dopamine receptor occupancy; antipsychotics; positron emission tomography
MeSH Terms: conditions — Schizophrenia | interventions — Positron-Emission Tomography; Mental Status and Dementia Tests; Therapeutics; Amisulpride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient group (Experimental): * 50 Drug-naïve patients with first episode psychosis (We anticipate the non-responder rate will be 30% of the patients)
    1. Drug-naïve
    2. Diagnosed as first episode psychosis
    3. The total score of PANSS>70
    4. No co-morbid psychiatric illness (including drug dependence/abuse)
  * They will also undergo PET scan at the baseline. And the investigators are going to determine treatment response after 6 weeks of treatment with amisulpride. Also they should complete clinical scales at 0, 2, 4, 6, and 8 week.
  Interventions: Device: PET scan; Behavioral: clinical scale; Drug: 6 weeks of treatment with amisulpride
- healthy control group (Other): * 12 healthy volunteers
    1. No history of psychiatric disorder (including drug dependence/abuse)
    2. No history of physical illness
    3. No contra-indication to scanning
  * They will also undergo PET scan at the baseline
  Interventions: Device: PET scan

INTERVENTIONS:
Device: PET scan — The patient group and the healthy control group will undergo PET scan at the baseline. the investigators are going to measure striatal dopamine synthesis capacity using [18 fluorine(F)]DOPA positron emission tomography in drug-naïve first episode psychosis and determine treatment response after 6 weeks of treatment with amisulpride. Response will be defined as a >30% reduction in symptom ratings on the Positive and Negative Syndrome Scale.
Behavioral: clinical scale — Patient group should complete clinical scales at baseline and 6 week.
  Arms: patient group
Drug: 6 weeks of treatment with amisulpride — The investigators are going to measure striatal dopamine synthesis capacity using [18 fluorine(F)]DOPA positron emission tomography in drug-naïve first episode psychosis and determine treatment response after 6 weeks of treatment with amisulpride. Response will be defined as a >30% reduction in symptom ratings on the Positive and Negative Syndrome Scale.
  Other Names: amisulpride
  Arms: patient group

SUMMARY:
The first purpose of this study is to determine if dopamine synthesis capacity is significantly lower in treatment non-responders from illness onset relative to treatment responders. And the second purpose of this study is to determine the potential of [18 fluorine(F)]-DOPA to be used to predict treatment response to antipsychotic treatment in first episode psychosis.

DETAILED DESCRIPTION:
Schizophrenia is amongst the leading causes of global disability in adults. A major factor underlying this is that about 30% of patients show little or no response to first-line antipsychotic drugs. There is one drug, clozapine, with proven efficacy in these patients. However, currently there are no good predictors of treatment non-response and consequently patients have to undergo empirical trials with first-line drugs. This contributes to the long delays, on average 4-5 years, seen in identifying and starting patients on clozapine. Furthermore, clozapine is poorly tolerated and has potentially life-threatening side-effects, which mean that the investigators desperately need new, alternative drugs. Lack of understanding of the neurobiological basis underlying non-response has impeded the development of alternatives to clozapine in the past. However recently it has been shown that non-responders show reduced dopamine synthesis capacity relative to patients who have responded to antipsychotics. The effect size for this difference is very large, d>1.2. This study was cross-sectional, in patients who had already received antipsychotic treatment for a number of years. The key questions now are thus:

1. is dopamine synthesis capacity different at illness onset in drug naïve patients who subsequently show non-response to antipsychotic treatment relative to drug naïve patients who respond to treatment
2. is it possible to predict who will respond to treatment

To test this the investigators are going to investigate the relationship between presynaptic dopamine dysfunction and antipsychotic responsiveness in a prospective study.

For this, the investigators are going to measure striatal dopamine synthesis capacity using [18 fluorine(F)]DOPA positron emission tomography in drug-naïve first episode psychosis and determine treatment response after 6 weeks of treatment with amisulpride. Response will be defined as a >30% reduction in symptom ratings on the Positive and Negative Syndrome Scale.

The effect size in our cross-sectional study was d=1.3. Based on this effect size a sample size of 12 per group will have >80% power to detect a group difference with p<0.05 2-tailed using an independent t-test. Given a non-response rate of 30% the investigators will thus require 40 patients at baseline to get 12 non-responders. To allow for 20% drop-outs we will require 50 patients at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Patient group (1) Patients who met Diagnostic and Statistical Manual of Mental Disorders(DSM)-IV criteria for schizophrenia, schizoaffective disorder, and schizophreniform disorder (2) Patients diagnosed with first episode psychosis which occurred within 2 years and not having been treated with antipsychotics(Drug-naïve) (3) The total score of PANSS>70
2. Healthy control group (1) Healthy controls has no Axis I disorder and do not report any past event of neurological or psychiatric illness assessed by the Structured Clinical Interview for DSM Disorders (2) No history of physical illness (3) No contra-indication to scanning

Exclusion Criteria:

1. Participants should not have any neurological illness such as head trauma, seizure and meningitis.
2. Participants should not be diagnosed as Mental retardation(IQ<70)
3. Participants should not have severe personality disorder, substance abuse or dependence (except for nicotine abuse and dependence) and severe medical conditions.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the difference of Ki(cer) of [18 fluorine(F)]DOPA PET | the difference of Ki(cer) between healthy controls and patient group at the baseline
  Subjects in the patient group will receive a intake of antipsychotics(amisulpride) for the six-week period and they will also undergo PET imaging at the baseline. After six-week marks, the investigators will determine treatment responders and nonresponders. And the investigators will detect the correlation between the capacity of presynaptic dopamine, treatment response and nonresponse in the patients.

SECONDARY OUTCOMES:
clinical scale(Positive and Negative Syndrome Scale) | change from baseline Positive and Negative Syndrome Scale and at 6 wk
  The investigators are going to measure striatal dopamine synthesis capacity using [18 fluorine(F)]DOPA positron emission tomography in drug-naïve first episode psychosis and determine treatment response after 6 weeks of treatment with amisulpride. Response will be defined as a >30% reduction in symptom ratings on the Positive and Negative Syndrome Scale.
Age | at baseline
  The investigators should check up participants' age
Sex | at baseline
  The investigators should check up participants' sex

CONTACTS AND LOCATIONS:
Overall Officials: Euitae Kim, Ph. D., Study Chair — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam

IPD SHARING:
Plan to Share IPD: Undecided